CLINICAL TRIAL: NCT04489329
Title: Use of the Small Intestine Microbiome Aspiration (SIMBA) Capsule to Detect a Dietary Intervention in the Small Intestine
Brief Title: Dietary Intervention Detection in the Small Intestine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nimble Science Ltd. (Industry)
Collaborators: University of Calgary (Other); Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REB 20-1211
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Proof of Concept
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Participant swallows and retrieves capsule in stool before and after ingestion of a probiotic. Capsule and stool samples are analyzed for presence of probiotic strain and compared to baseline.
  Interventions: Device: Ingestible Capsule; Dietary Supplement: Probiotic

INTERVENTIONS:
Device: Ingestible Capsule — Participants will swallow capsule and undergo X-rays to establish transit
Dietary Supplement: Probiotic — Participants will swallow a probiotic capsule and the sample collection capsule at the same time to establish concentration of strain in small intestine.

SUMMARY:
Proof of concept study to validate the ability of a capsule device to gather samples from the small bowel for microbiome analysis in adults and to detect dietary changes from simultaneous ingestion of a probiotic.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old
2. Healthy
3. On no medication, or on stable doses of medications which will not be changed over the course of the study
4. Willingness to maintain their usual dietary habits and physical activity
5. Willing to discontinue consumption of fermented foods or probiotics (such as kombucha, yogurts with live, active cultures, or probiotic supplements) for the duration of the study.
6. Ability to understand and provide informed consent
7. Ability and willingness to meet the required schedule and study tasks and interventions
8. Willing to fast for at least 8 hours before the 2 intake visits (Visit 1 and Visit 2)

Exclusion Criteria:

1. History of a small intestine obstruction of symptoms of an intermittent small intestine obstruction (i.e., recurrent abdominal pain, distention, nausea and vomiting).
2. Pregnant or breastfeeding or planning on becoming pregnant during study timeline.
3. Use of other investigational product within 3 months of start of the study.
4. Suffering from immune disorders or with possible immune deficient status
5. Allergy to soy or milk.
6. Prior gastrointestinal surgery which has altered the anatomy of the esophagus, stomach or small or large intestine (exceptions include appendectomy or cholecystectomy more than 3 months prior to enrollment).
7. Use of any medications in the previous 7 days that could substantially alter gastrointestinal motor function (e.g. opioids, prokinetics, anticholinergics, laxatives), acidity (PPI, H2RA), or integrity (NSAIDs, oral steroids).
8. Body Mass Index (BMI) > 38.
9. Previous history of gastric bezoar or gastroparesis.
10. Any abdominal or pelvic surgery within the past 3 months.
11. Known history of inflammatory bowel disease and/or Crohn's disease.
12. History of diverticulitis, diverticular stricture, or other intestinal strictures.
13. History of abdominal or pelvic radiotherapy.
14. History of dysphagia, eosinophilic esophagitis, esophageal stricture, or other swallowing disorder.
15. Cardiovascular, endocrine, renal or other chronic disease likely to affect motility.
16. Colon cleansing prep for 1 month before the first visit, or during the study.
17. Use of antibiotics, prebiotics, herbal supplements, or probiotics for 2 weeks before the first visit, or during the study.
18. < 2 bowel movements per week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Bacterial density count | 7 days
  density count of probiotic strain compared between capsule and stool sample (CFU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Andrews, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- Cumming School of Medicine, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No